CLINICAL TRIAL: NCT05346237
Title: Validation and Cross-cultural Adaptation of Croatian Self-Evaluation of Communication Experiences After Laryngectomy Questionnaire
Brief Title: Validation and Cross-cultural Adaptation of Croatian SECEL Questionnaire
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OsijekUH-SECEL
Record Dates: First submitted 2022-04-13; First posted 2022-04-26 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: Larynx Neoplasm; Laryngectomy; Status; Communication; Quality of Life
Keywords: Laryngectomy; Speech,alaryngeal; Quality of Life; Assessment; Communication
MeSH Terms: conditions — Laryngeal Neoplasms; Communication; Speech

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult laryngectomised patients: Patients who have undergone total laryngectomy and completed minimal their 12-month period without disease after surgery and post-operative treatments such as radiotherapy or chemotherapy
  Interventions: Behavioral: Quality of life questionnaire

INTERVENTIONS:
Behavioral: Quality of life questionnaire — Filling out questionnaires, measuring maximum phonation and diadochokinesis

SUMMARY:
Self-Evaluation of Communication Experiences after Laryngectomy (SECEL) questionnaire has been developed, with the aim of evaluating rehabilitation needs and the psychosocial care for patients with laryngeal cancer. This short but comprehensive self-report instrument measures the perceived adjustment to communication experiences and is intended to aid in determining counselling needs in patients with laryngeal cancer who are treated with a laryngectomy. The first aim of this study is to evaluate the translation, psychometric properties and cultural adaptation of a Croatian version of the SECEL questionnaire. Secondary aim is to examine relationship between the Croatian version of the SECEL and the Short Form Health Survey (SF-36) and the Voice Handicap Index (VHI) questionnaires and to examine relationship between objective voice measures and Self-Evaluation of Communication Experiences after Laryngectomy (SECEL:HR).

DETAILED DESCRIPTION:
At the first visit all patients included in the study were asked to complete the Croatian version of the Voice Handicap Index (VHI), Short Form Health Survey (SF-36) and Self-Evaluation of Communication Experiences after Laryngectomy (SECEL:HR) questionnaire.

SECEL questionnaire consists of two parts. The first part examines the relevant general data on the person filling out the questionnaire, while the second part consists of 35 items questionably or statement-designed to examine communication experiences. Patients estimates the incidence of these communication difficulties on the Likert scale (0-never, 1-sometimes, 2-often, 3-always). 35 items are grouped according to 3 subscales named General (0-15 score range), Environment (0-42 score range) and Attitude (0-45 score range), and item number 35 is a separate question: "Do you talk the same amount now as before your laryngectomy?" and is rated with a "yes," "more," and "less" rating category. The overall numerical score varies from 0 to 102, and the higher score indicates greater difficulties and worse postoperative speech-communication adjustment.

The Voice Handicap Index (VHI) questionnaire consist of 30 items organized in three subscales functional, physical and emotional and also scored with Likert scale with overall score from 0 to 120. Higher scores indicate a greater handicap.

The Short Form Health Survey (SF-36) is a multi-purpose short-form health survey that consist of 36 questions divided in eight dimension and clustered into two groups: physical and mental health. Each item was standardized (range 0-100), with a higher score representing better QoL.

The objective assessment includes the maximum phonation time measured in seconds as common clinical measure of glottal efficiency, diadochokinesis of the 3-syllable "pa-ta-ka" in 5 seconds (rated in syll/s) or how quickly subjects can produce a series of rapid sounds which is a measure of speech efficiency.

All patients will fulfil the SECEL:HR questionnaire twice, two weeks after the initial test and that will be considered as a re-test of the SECEL reliability analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed minimal their 12-month period without disease after surgery and post-operative treatments such as radiotherapy or chemotherapy
2. Patients with preserved reading skills
3. Regular presence at follow-up visits

Exclusion Criteria:

1. Acute respiratory infection of the upper or lower respiratory tract
2. Presence of neurologic or pulmonary diseases
3. Recurrence of cancer
4. Deviation from the research protocol

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who have undergone total laryngectomy were included in this study
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Željka Laksar Klarić, M.D., Principal Investigator — Clinical Department of ENT and Head and Neck Surgery, Clinical Hospital Centre Osijek
Locations (1):
- University Hospital Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schindler A, Mozzanica F, Brignoli F, Maruzzi P, Evitts P, Ottaviani F. Reliability and validity of the Italian self-evaluation of communication experiences after laryngeal cancer questionnaire. Head Neck. 2013 Nov;35(11):1606-15. doi: 10.1002/hed.23198. Epub 2012 Nov 20. PMID 23169480
- [Background] Finizia C, Bergman B, Lindstrom J. A cross-sectional validation study of Self-Evaluation of Communication Experiences after Laryngeal Cancer--a questionnaire for use in the voice rehabilitation of laryngeal cancer patients. Acta Oncol. 1999;38(5):573-80. doi: 10.1080/028418699431159. PMID 10427945
- [Background] Lundstrom E, Hammarberg B. Speech and voice after laryngectomy: perceptual and acoustical analyses of tracheoesophageal speech related to voice handicap index. Folia Phoniatr Logop. 2011;63(2):98-108. doi: 10.1159/000319740. Epub 2010 Oct 8. PMID 20938189
- [Background] Johansson M, Ryden A, Finizia C. Self evaluation of communication experiences after laryngeal cancer - a longitudinal questionnaire study in patients with laryngeal cancer. BMC Cancer. 2008 Mar 27;8:80. doi: 10.1186/1471-2407-8-80. PMID 18371189
- [Background] Bonetti A, Bonetti L. Cross-cultural adaptation and validation of the Voice Handicap Index into Croatian. J Voice. 2013 Jan;27(1):130.e7-130.e14. doi: 10.1016/j.jvoice.2012.07.006. Epub 2012 Oct 6. PMID 23044461
- [Background] Maslic Sersic D, Vuletic G. Psychometric evaluation and establishing norms of Croatian SF-36 health survey: framework for subjective health research. Croat Med J. 2006 Feb;47(1):95-102. PMID 16489702
- [Derived] Laksar Klaric Z, Danic Hadzibegovic A, Vceva A, Karadza Lapic L, Babler D, Kralik K, Bonetti A, Bensic A. Validation and Cross-Cultural Adaptation of Croatian Self-Evaluation of Communication Experiences after Laryngectomy Questionnaire. Folia Phoniatr Logop. 2023;75(5):273-283. doi: 10.1159/000529771. Epub 2023 Feb 17. PMID 36808105

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adult Laryngectomised Patients
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Laryngectomised Patients
Number analyzed (Participants) | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [63 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Tumor stage [Count of Participants; unit: Participants] — Tumor stage -primary tumor T1 - the tumor is limited to the vocal cords with normal mobility T2 - the tumor spreads to the supraglottis and/or subglottis or a tumor with limited mobility of the vocal cords T3 - the tumor is confined to the larynx with fixation of the vocal cords T4- the tumor invades the thyroid or cricoid cartilage or affects tissue outside the larynx
  Participants
    T1- affects a vocal cord with neck metastases in ipsilateral nodes that are no larger than 6 cm | 1
    T2 | 9
    T3 | 21
    T4 | 17
Smoking habits [Count of Participants; unit: Participants]
  Never smokers | 3
  Smokers | 2
  Ex-smokers | 45
Time since surgery [Count of Participants; unit: Participants]
  12-24 months | 12
  > 24 months | 38
Radiotherapy [Count of Participants; unit: Participants]
  No | 18
  Before surgery | 1
  After surgery | 31
Chemotherapy [Count of Participants; unit: Participants] | 18
Education completed [Count of Participants; unit: Participants]
  Elementary school | 16
  High school | 29
  Undergraduate studies | 3
  Graduate studies | 1
  Post-graduate studies | 1

OUTCOME MEASURES:

1. Primary Outcome: Means, Standard Deviations (Ranges), Test-retest Reliability of the Self- Evaluation of Communication Experiences After Laryngectomy (SECEL:HR) Questionnaire
Description: Completing the Croatian version of the SECEL questionnaire. Questionnaire consists of two parts. The first part examines the relevant general data on the person filling out the questionnaire, while the second part consists of 35 items questionably or statement-designed to examine communication experiences. Patients estimates the incidence of these communication difficulties on a 4-point scale (0-never, 1-sometimes, 2-often, 3-always) The 35 items are grouped according to 3 subscales named General (0-15 score range), Environment (0-42 score range) and Attitude (0-45 score range). Item number 35 is a separate question: "Do you talk the same amount now as before your laryngectomy?" and is rated with a "yes," "more," and "less" rating category. The overall numerical score varies from 0 to 102, where the higher score indicates greater difficulties and worse postoperative speech-communication adjustment.
Time Frame: 15 minutes- required to complete the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SECEL:HR = General Subscale: General subscale - questions or statements, intended to examine communication experiences. Patients estimate the incidence of these communication difficulties on the Likert scale (0-never, 1-sometimes, 2-often, 3-always). General (0-15 score range),
- SECEL:HR = Environment Subscale: Environment subscale - questions or statements, intended to examine communication experiences. Patients estimate the incidence of these communication difficulties on the Likert scale (0-never, 1-sometimes, 2-often, 3-always). Environment subscale (0-42 score range).
- SECEL:HR = Attitude Subscale: Attitude subscale - questions or statements, intended to examine communication experiences. Patients estimate the incidence of these communication difficulties on the Likert scale (0-never, 1-sometimes, 2-often, 3-always). Attitude subscale (0-45 score range)
- SECEL:HR = Total: 35 items designed as questions or statements and intended to examine communication experiences. Patients estimate the incidence of these communication difficulties on the Likert scale (0-never, 1-sometimes, 2-often, 3-always). The 35 items are grouped according to 3 subscales named General (0-15 score range), Environment (0-42 score range) and Attitude (0-45 score range)
Arm/Group | SECEL:HR = General Subscale | SECEL:HR = Environment Subscale | SECEL:HR = Attitude Subscale | SECEL:HR = Total
Number analyzed (Participants) | 50 | 50 | 50 | 50
units on a scale
  Re- Test (standard deviation) | 4.69 (2.7) | 16.33 (8.4) | 9.38 (8.8) | 30.10 (17.5)
  Test (standard deviation) | 4.21 (2.4) | 14.85 (2.4) | 7.49 (7.0) | 26.51 (14.1)

2. Primary Outcome: Means, Standard Deviations of SF-36
Description: Completing the Croatian version of the Short Form Health Survey (SF-36) questionnaire. The SF-36 consist of 36 questions divided in eight dimension and clustered into two groups: physical and mental health. The 8 groups of questions are: physical functioning (SF-PF), role limitations due to physical problems (SF-RP), bodily pain ( SF-BP), general health (SF-GH), vitality (SF-VT), social functioning (SF-SF), emotional role ( SF-RE), mental health (SF-MH), change in health (SF-HC).
  To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Time Frame: 15 minutes- required to complete the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SF-PF; SF-VT: Range 35-100
  (to score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software)
- SF-RP; SF-RE: Range 0-100
  (to score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software)
- SF-BP: Range 10-100
  (to score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software)
- SF-GH: Range 30-100
  (to score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software)
- SF-SF: Range 38-100
  (to score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software)
- SF-MH: Range 36-100
  (to score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software)
- SF-HC: Range 25-100
  (to score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software)
Arm/Group | SF-PF | SF-RP | SF-BP | SF-GH | SF-VT | SF-SF | SF-RE | SF-MH | SF-HC
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50 | 50 | 50 | 50
units on a scale | 75.50 (16.2) | 60.00 (41.3) | 77.20 (26.1) | 62.60 (15.8) | 68.20 (18.2) | 78.38 (20.6) | 78.02 (37.9) | 72.88 (19.6) | 56.00 (22.3)

3. Primary Outcome: Means, Standard Deviation of VHI Questionnaire
Description: Completing the Croatian version of the Voice Handicap Index (VHI) questionnaire. The Voice Handicap Index (VHI) questionnaire consist of 30 items organized in three subscales: functional, physical and emotional, scored on 5-point scale (0-never, 1-almost never, 2-sometimes, 3-almost always, 4-always) with overall score from 0 to 120. Higher scores indicate a greater handicap.
Time Frame: 15 minutes-required to complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- VHI E - Emotional Subscale of VHI; VHI F- Functional Subscale of VHI; VHI P - Physical Subscale of VHI: scored on 5-point scale (0-never, 1-almost never, 2-sometimes, 3-almost always, 4-always)
- VHI TOT - VHI Total Score: scored on 5-point scale (0-never, 1-almost never, 2-sometimes, 3-almost always, 4-always).
  Overall score from 0 to 120. Higher scores indicate a greater handicap.
Arm/Group | VHI E - Emotional Subscale of VHI | VHI F- Functional Subscale of VHI | VHI P - Physical Subscale of VHI | VHI TOT - VHI Total Score
Number analyzed (Participants) | 50 | 50 | 50 | 50
score on a scale | 7.50 (7.6) | 15.84 (7.6) | 12.70 (8.7) | 35.86 (19.9)

4. Secondary Outcome: Mean, Standard Deviation of Maximum Phonation Time (MPT) and Diadochokinesis (DDK)
Description: The maximum phonation time (measured in seconds) for which a person can sustain a vowel sound when produced on 1 deep breath at a comfortable pitch and loudness and is a common clinical measure of glottal efficiency.
  Diadochokinesis of the 3-syllable "pa-ta-ka" in 5 seconds (rated in syll/s),and the number of syllables per second of the 5 sentences. Diadochokinesis measures how quickly an individual can accurately produce a series of rapid, alternating sounds and is a simple and common clinical measure of speech efficiency.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: mesured in seconds
Groups:
- MPT - The Maximum Phonation Time: The maximum phonation time (measured in seconds) for which a person can sustain a vowel sound when produced on 1 deep breath at a comfortable pitch and loudness and is a common clinical measure of glottal efficiency.
- DDK -Diadochokinesis: Diadochokinesis of the 3-syllable "pa-ta-ka" in 5 seconds (rated in syll/s),and the number of syllables per second of the 5 sentences. Diadochokinesis measures how quickly an individual can accurately produce a series of rapid, alternating sounds and is a simple and common clinical measure of speech efficiency.
Arm/Group | MPT - The Maximum Phonation Time | DDK -Diadochokinesis
Number analyzed (Participants) | 50 | 50
mesured in seconds | 8.55 (4.2) | 8.94 (2.0)

ADVERSE EVENTS:
Time Frame: 15 minutes
Description: The SECEL is a 35-item patient-reported questionnaire developed to address the communication needs of patients with laryngectomies. The aim was to translate, cross-culturally adapt and validate Croatian version. The SECEL:HR was filled in by 50 laryngectomised patients.
Arm/Group | Adult Laryngectomised Patients
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT05346237/Prot_SAP_002.pdf